CLINICAL TRIAL: NCT00485121
Title: Effects of Ezetimibe Add-On to Statin Therapy on Adipokine Production in Obese and Metabolic Syndrome Patients With Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Collaborative Research Network (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05080
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Syndrome; Obesity; Coronary Artery Disease
Keywords: Ezetimibe; Statin; Low- density lipoprotein cholesterol; Adipokine; Adiponectin; C-reactive protein; Coronary artery disease; Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Coronary Artery Disease | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ezetimibe

SUMMARY:
The purpose of this study is to investigate the effects of adding ezetimibe to statin therapy on levels of inflammatory markers and adipokines in patients with atherosclerosis disease and features of the metabolic syndrome,whose LDL-c remains above target (> 2.0 mmol/L) despite statin monotherapy.

We hypothesize that the addition of Ezetimibe (10mg per day for 12 weeks) to ongoing statin therapy in patients with atherosclerosis and features of the metabolic syndrome will favourably modify levels of inflammatory biomarkers and adipokines.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease remains the leading cause of death in industrialized nations despite major advances in its diagnosis, treatment and prevention. While there has been a trend over the last half century showing a general decline in the age-adjusted death rates of heart disease and stroke, the increasing epidemic of obesity, followed closely by insulin resistance and type 2 diabetes will likely slow the decline and promise to reverse this trend.

Obesity mediates increased cardiovascular disease risks through multiple pathways. Adipose tissue is no longer viewed as a passive repository for triacylglycerol storage and a source of free fatty acids (FFAs). It is recognized as a rich source of proinflammatory mediators, many of which are cytokines, growth factors and hormones that directly contribute to the proinflammatory milieu mediating vascular injury, insulin resistance and ultimately impacting on cardiovascular health. These proinflammatory adipocytokines, or adipokines include tumor necrosis factor- α (TNF α), interleukin-6 (IL-6), leptin, plasminogen activator inhibitor-1 (PAI-1), angiotensinogen, resistin and more recently C-reactive protein (CRP). On the other hand, nitric oxide (NO) and another adipokine called adiponectin confer protection against inflammation and obesity-linked insulin resistance.

The evolving role of augmented adipokine production in obese and insulin resistant states in cardiovascular disease risk opens new avenues for therapeutic interventions. Treatment of the metabolic syndrome will need to embrace new strategies to reduce the burden of proinflammatory adipokines. Lifestyle intervention remains the cornerstone therapy, but considerations should also be given to a number of drugs that can decrease the inflammatory adipokines.

Ezetimibe selectively inhibits the absorption of biliary and dietary cholesterol and phytosterols at the intestinal brush border. When added to or coadministered with a statin, ezetimibe produces significant incremental LDL-C, apolipoprotein (apo) B, and triglyceride (TG) reductions, beneficial effects on high-density lipoprotein cholesterol (HDL-C) compared to statin monotherapy, and is well tolerated with a low incidence of side effects.

It was previously demonstrated that in a 12 week trial that the addition of ezetimibe to simvastatin resulted in significant incremental reductions in CRP compared to simvastatin monotherapy.

The outlined study protocol investigates the effects of adding ezetimibe to statin therapy on levels of inflammatory markers and adipokines in patients with atherosclerosis and features of the metabolic syndrome, whose LDL-c remains above target (> 2.0 mmol/L) despite statin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients on statin therapy (no dose change within past 4 weeks) with LDL-c > 2mmol/l
* Presence of atherosclerosis (CHD* and/or cerebrovascular disease** and/ or peripheral arterial disease (PAD)***) plus at least one of the following:

  1. Metabolic Syndrome (according to modified NCEP ATP III criteria, using waist circumference cut-offs of 80 cm for women and 90 cm for men in all subjects of Asian origin and cut-offs of 88 cm for women and 102 cm for men in all Caucasian subjects)
  2. Obesity (BMI > 30 Kg/m2 or waist circumference of > 102 for men and > 88 for women. For subjects of Asian origin the cutoff values should be 25, 90 and 80 respectively)

     * CHD defined as (any one of the following): previous myocardial infarction; coronary angiography demonstrating at least 50% diameter stenosis in an epicardial coronary artery or its major branch; previous percutaneous transluminal coronary angioplasty (PTCA) with or without stent implantation (atherectomy included) or previous coronary artery bypass grafting (CABG)

       * Cerebrovascular disease defined as (any one of the following): prior ischemic stroke, documented TIA, or flow-limiting stenosis in extracranial artery documented by Doppler or angiography.

         * PAD defined as (any one of the following): prior peripheral arterial revascularization (PTA or surgery), amputation, or documented intermittent claudication with ABI < 0.9

Exclusion Criteria:

* Women who are pregnant, breast feeding, or not using a reliable method of contraception
* Clinical signs of congestive heart failure or measured left ventricular ejection fraction <40%
* Hemodynamically significant valvular heart disease or hypertrophic obstructive cardiomyopathy
* Renal dysfunction (creatinine > 1.8 x ULN)
* Hepatic disease (liver function test >1.5 x ULN [upper limit normal])
* Other significant laboratory abnormalities that the investigator feels may compromise the patient's safety by participation in the study
* History of systemic inflammatory disease (rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematous), myositis/myopathic process, or cancer)
* HIV
* Use of steroids or chemotherapy drugs within the past year or chronic use of nonsteroidal anti-inflammatory drugs besides aspirin (use for > 2 weeks within the past year);
* Known hypersensitivity to Ezetimibe
* Participation in another clinical study concurrently or within the 30-day phase prior to screening for entry into the present study
* Unwilling to provide written informed consent for study participant and/or
* Unreliability as a study participant as based on the investigator's prior knowledge of the patient, such as the inability or willingness to participate in or complete the study or the presence of concurrent physical or psychological disorders that may make it impractical for the patient to participate in or complete the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in adiponectin levels | 12 weeks

SECONDARY OUTCOMES:
Change in CRP, PAI-1, Il-6, TNF-α, resistin, leptin levels and serum lipids (total cholesterol, HDL-cholesterol, LDL-cholesterol, Triglycerides). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Milan K Gupta, MD, Principal Investigator — Partners Research
Locations (1):
- Partners Research, Brampton, Ontario, Canada